CLINICAL TRIAL: NCT05861791
Title: Comparison of Patient-controlled Analgesia With Background Opioid Versus Non-opioid Infusion for Postoperative Pain in Patients Undergoing Total Knee Arthroplasty: a Randomized, Non-inferiority Study
Brief Title: Comparison of Patient-controlled Analgesia Regimenfor Postoperative Pain in Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University Gwangmyeong Hospital (Other)
Responsible Party: Principal Investigator, Se-Hee Min, Assistant professor, Chung-Ang University Gwangmyeong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2210033049
Record Dates: First submitted 2023-02-08; First posted 2023-05-17 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Ketorolac Tromethamine; Nefopam

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid group (Experimental): IV-PCA consisted of fentanyl
  Interventions: Drug: Fentanyl
- non-opioid group (Active Comparator): IV-PCA consisted of ketorolac and nefopam
  Interventions: Drug: ketorolac tromethamine with nefopam hydrochloride

INTERVENTIONS:
Drug: Fentanyl — opioid group receives only fentanyl citrate 1200mcg for continuous infusion drug
  Other Names: opioid group
  Arms: opioid group
Drug: ketorolac tromethamine with nefopam hydrochloride — non-opioid group receives ketorolac tromethamine 150mg with nefopam hydrochloride 100mg for continuous infusion drug
  Arms: non-opioid group

SUMMARY:
Patients who undergoing total knee arthroplasty under spinal analgesia will be recruited and randomly assigned to the following two groups according to the regimen of PCA: (A) opioid group who receive only fentanyl citrate 1200mcg for continuous infusion drug, (B) non-opioid group who receive ketorolac tromethamine 150mg with nefopam hydrochloride 100mg for continuous infusion drug. All the patients will receive additional fentanyl citrate as bolus injection drug if they need more analgesics postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* undergoing elective total knee arthroplasty under spinal anesthesia

Exclusion Criteria:

* history of stomack ulceration
* increased ICP
* bronchial asthma
* allergy on aspirin, NSAIDs, Nefopam
* drug user of antiplatelet or anticoagulant

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
postoperative pain score | 24 hours after the surgery
  evaluated by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hee Min, Principal Investigator — ChungAng University Gwangmyeon Hospital
Locations (1):
- ChungAng University Gwangmyeong Hospital, Gyeonggi-do, Gwangmyeon-si, South Korea